CLINICAL TRIAL: NCT05620693
Title: Study NY-ESO-1 TCR-T in Advanced Soft Tissue Sarcoma
Brief Title: Study of NY-ESO-1 TCR-T in Advanced Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-022
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Advanced Soft-tissue Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): TCR-T treatment group
  Interventions: Biological: NY-ESO-1 TCR-T

INTERVENTIONS:
Biological: NY-ESO-1 TCR-T — NY-ESO-1 TCR-T treatment

SUMMARY:
Soft tissue sarcoma (STS) is a kind of solid tumor with high heterogeneity. There is no standard second-line treatment plan for patients who have failed first-line treatment. NY-ESO-1, a cancer testis antigen, is highly expressed in soft tissue tumors and is an ideal therapeutic target.

Investigators aim to testify the safety and efficacy of NY-ESO-1 TCR-T cell in advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
Soft tissue sarcoma (STS) is a kind of solid tumor with high heterogeneity. The treatment of STS is complex and challenging, and surgery is still the main treatment method at present. For patients who are inoperable or advanced, medical treatment should be considered, mainly including chemotherapy and targeted treatment. At present, there is no standard second-line treatment plan for patients who failed first-line treatment.

NY-ESO-1, a cancer testis antigen, is highly expressed in soft tissue tumors and is an ideal therapeutic target.

Investigators aim to testify the safety and efficacy of NY-ESO-1 TCR-T cell in advanced soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 (≥ 18, ≤ 70), regardless of gender;
2. Subjects voluntarily participate in the study, and they or their legal guardians sign the Informed Consent Form;
3. Late recurrent or metastatic soft tissue sarcoma confirmed by histopathology; Progress after receiving first-line treatment;
4. According to RECIST 1.1 standard, there are clear assessable lesions;
5. The expression of NY-ESO-1 in tumor tissue was confirmed by immunohistochemical staining; HLA-A configuration is 02/01;
6. Within 2 weeks before cell therapy, no antibody drugs were used;
7. ECOG score is 0-2;
8. The subject has no contraindication for peripheral blood collection;
9. The expected survival period is more than 3 months.

Exclusion Criteria:

1. People who have a history of allergy to any component in cell products;
2. The following conditions occur in blood routine examination: WBC ≤ 1 × 109/L, absolute value of neutrophil ANC ≤ 0.5 × 109/L, absolute value of lymphocyte ALC ≤ 0.5 × 109/L , PLT≦25 × 109/L ；
3. The following conditions occur in laboratory testing: including but not limited to, total serum bilirubin ≥ 1.5mg/dl; Serum ALT or AST is more than 2.5 times of the upper limit of normal; Blood creatinine ≥ 2.0mg/dl;
4. According to the NYHA cardiac function grading standard, patients with cardiac insufficiency belong to Grade III or IV; Or left ventricular ejection fraction (LVEF)<50% by echocardiography;
5. Pulmonary function is abnormal, and the saturation of blood oxygen under indoor air is less than 92%;
6. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other serious heart diseases clinically within 12 months before enrollment;
7. Grade 3 hypertension and poor blood pressure control after drug treatment;
8. Have suffered from brain trauma, consciousness disorder, epilepsy, relatively serious cerebral ischemia or cerebral hemorrhage disease in the past;
9. Patients with autoimmune diseases, immunodeficiency or other patients requiring immunosuppressive treatment;
10. There is uncontrolled active infection;
11. Have used any cell therapy products in recent 3 months;
12. Live vaccine inoculation within 4 weeks before enrollment;
13. HIV, HBV, HCV and TPPA/RPR positive persons, and HBV carriers;
14. Subjects have a history of alcohol abuse, drug abuse or mental illness;
15. Subjects have participated in any other clinical research within 3 months before joining this clinical research;
16. Female subjects have any of the following conditions: a) are in pregnancy/lactation; Or b) having a pregnancy plan during the trial; Or c) is fertile and unable to take effective contraceptive measures;
17. The investigator believes that there are other circumstances that are not suitable for the subject to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
AE/SAE | from infusion to 30 days after infusion
  adverse events/ sever adverse events

SECONDARY OUTCOMES:
ORR | From admission to the end of follow up, up to 2 years.
  overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No